CLINICAL TRIAL: NCT01182909
Title: Far Eastern Memorial Hospital
Brief Title: Environmental and Genetic Determinants of Nasopharyngeal Carcinoma (NPC)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Collaborators: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, Li-Jen Liao, Department of Otolaryngology, Far Eastern Memorial Hospital
Other Study IDs: 099046-F
Record Dates: First submitted 2010-08-15; First posted 2010-08-17 (Estimated); Last update posted 2011-09-19 (Estimated); Status verified 2011-09

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: NPC; Environmental and Genetic; evaluate putative environmental exposures and NPC; assess the effect of genetic factors; investigate gene-environment interactions; examine the natural history of EBV infection
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Nasopharyngeal carcinoma (NPC) is one of the most common malignant tumors in southern China and Southeast Asia. While infection with Epstein-Barr Virus (EBV) is believed to be necessary for the development of NPC, non-viral environmental factors have also been implicated to increase the risk of NPC including consumption of salted fish and other nitrosamine containing preserved foods, formaldehyde and wood dust exposure, and cigarette smoking. In addition to environmental factors, it is widely accepted that genetic susceptibility also plays an important role in the pathogenesis of NPC. Polymorphisms in genes involved in nitrosamine metabolism and DNA repair have been suggested to be associated with NPC risk, and various chromosomal regions linked to NPC development have been reported. These associations highlight the role of both environmental and genomic components in the etiology of NPC.

There is a longstanding history of international collaborative studies to elucidate the role of environmental and genetic factors associated with NPC between investigators in Taiwan and the USA. A case-control study (375 cases; 327 controls) was conducted in the early 1990s, and a large multiplex family study that was completed in 2006 (358 families; 3,216 individuals). Results from these studies have provided some of the most comprehensive epidemiological evidence regarding factors linked to NPC development to date.

As a next logical step, the opportunity now exists to undertake a genome-wide association study of NPC in Taiwan with carefully collected environmental exposure data to systematically examine environmental and genetic factors associated with NPC, and to evaluate gene-gene and gene-environment interactions. The investigators propose a case-control study of 2000 NPC cases (both retrospective [n=800] and prospective [n=1,200]) and 2,000 age-gender-matched hospital controls in northern Taiwan. The study objectives are to: 1) evaluate putative environmental exposures and NPC; 2) assess the effect of genetic factors, including both single nucleotide polymorphism and copy number variation through analysis of both main effect and gene-gene interaction; 3) investigate gene-environment interactions by testing for interactions between significant genome-wide genetic variations and EBV and other identified environmental risk factors; and 4) examine the natural history of EBV infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with NPC

Exclusion Criteria:

* Case group and control group younger than 18 age. Control group, the reasons for hospitalization for the EB virus-related disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We propose a case-control study of 2000 NPC cases (both retrospective [n=800] and prospective [n=1,200]) and 2,000 age-gender-matched hospital controls in northern Taiwan
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2010-08; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, Taipei, Taiwan